CLINICAL TRIAL: NCT00102739
Title: See Detailed Description
Brief Title: SB-497115 (Oral Thrombopoietin Receptor Agonist) Versus Placebo In Adults With Refractory Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRA100773
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2012-11

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: thrombopoietin; immune thrombocytopenic purpura; platelets; chronic thrombocytopenia
MeSH Terms: conditions — Purpura; Jacobs syndrome; Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB497115

SUMMARY:
This study is a double-blind, randomized, placebo-controlled, parallel group, repeat-dose, study conducted in two parts (Part A and Part B) examining 30, 50, and 75 mg doses of SB-497115-GR as a treatment for patients with ITP who have failed prior therapy. The study is designed to determine the proportion of patients with a platelet count =50,000/µL after 42 days. In Part B, 99 newly-recruited subjects will be randomized to one of two dosing arms in a 2:1 ratio of active:placebo. During the 6 week study period, subjects will start on placebo or active drug (50 mg) and may have a dose increase to 75 mg based upon their platelet count at day 22.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, parallel group study to investigate the efficacy, safety, tolerability, pharmacokinetics, and pharmacodynamics of SB-497119-GR, a thrombopoietin receptor agonist, administered at 30, 50, and 75 mg as oral tablets once-daily for 6 weeks to adult male and female subjects with refractory, chronic immune thrombocytopenia purpura

ELIGIBILITY:
Inclusion criteria:

* Patients with chronic low platelet count (less than 30,000/µL) for 6 months who have failed at least one treatment for chronic low platelet count.
* Patients receiving chronic maintenance steroid therapy must have received a stable dose for at least 1 month.
* Normal PT and PTT.

Exclusion criteria:

* History of clotting disorder.
* Females who are pregnant or are receiving hormone replacement therapy or systemic contraceptives.
* History of alcohol/drug abuse or dependence within 1 year.
* Use of aspirin, aspirin-containing compounds, salicylates, antacids, rosuvastatin, pravastatin, non-steroidal anti-inflammatory drugs during the study and within 3 weeks prior to starting the study.
* History of HIV infection or active infection with Hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Treatment response, assessed by the proportion of patients with platelet counts of =50, 000/µL (compared with baseline count of <30, 000/µL) after 42 days of treatment.

SECONDARY OUTCOMES:
Safety, tolerability, PK, PD, symptoms associated with ITP, and QoL, odds of response vs placebo during weeks 2 to 6 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- GSK Investigational Site, Bad Nauheim, Hesse, Germany
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- GSK Investigational Site, Auckland, New Zealand
- GSK Investigational Site, Lahore, Pakistan
- GSK Investigational Site, Lodz, Poland
- GSK Investigational Site, Bucharest, Romania
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
- Slovenia (2):
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Maribor
- GSK Investigational Site, Seoul, South Korea
- GSK Investigational Site, Taipei, Taiwan
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
- United Kingdom (6):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Taunton, Somerset
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Swansea

REFERENCES:
- [Background] Bussel JB, Cheng G, Saleh MN, Psaila B, Kovaleva L, Meddeb B, Kloczko J, Hassani H, Mayer B, Stone NL, Arning M, Provan D, Jenkins JM. Eltrombopag for the treatment of chronic idiopathic thrombocytopenic purpura. N Engl J Med. 2007 Nov 29;357(22):2237-47. doi: 10.1056/NEJMoa073275. PMID 18046028
- [Background] Gibiansky E, Zhang J, Williams D, Wang Z, Ouellet D. Population pharmacokinetics of eltrombopag in healthy subjects and patients with chronic idiopathic thrombocytopenic purpura. J Clin Pharmacol. 2011 Jun;51(6):842-56. doi: 10.1177/0091270010375427. Epub 2010 Jul 27. PMID 20663993
- [Derived] Tarantino MD, Fogarty P, Mayer B, Vasey SY, Brainsky A. Efficacy of eltrombopag in management of bleeding symptoms associated with chronic immune thrombocytopenia. Blood Coagul Fibrinolysis. 2013 Apr;24(3):284-96. doi: 10.1097/MBC.0b013e32835fac99. PMID 23492914
- [Derived] Bussel JB, Provan D, Shamsi T, Cheng G, Psaila B, Kovaleva L, Salama A, Jenkins JM, Roychowdhury D, Mayer B, Stone N, Arning M. Effect of eltrombopag on platelet counts and bleeding during treatment of chronic idiopathic thrombocytopenic purpura: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Feb 21;373(9664):641-8. doi: 10.1016/S0140-6736(09)60402-5. PMID 19231632